CLINICAL TRIAL: NCT00512863
Title: A Phase 2a, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel, Dose-Finding Study to Evaluate the Safety, Efficacy and Pharmacokinetics of Adalimumab in Subjects With Refractory Asthma
Brief Title: A Dose-Finding Study to Evaluate the Safety, Efficacy and Pharmacokinetics of Adalimumab in Subjects With Refractory Asthma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M05-757
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Last update posted 2007-11-06 (Estimated); Status verified 2007-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Humira (adalimumab)

SUMMARY:
To evaluate the efficacy of SC injections of 3 regimens of adalimumab vs. placebo in the change in post-bronchodilator FEV1 from Baseline to Week 16 when used in the treatment of refractory asthma.

ELIGIBILITY:
Inclusion Criteria:

* Documented history of refractory asthma, as defined by the American Thoracic Society,31 defined as 1 major and at least 2 minor criteria
* Actual or documented history of reversible airway obstruction
* Baseline FEV1 of 40% - 80% of the predicted for height, age, and sex at Screening, as demonstrated 6 or more hours after a short-acting -agonist and/or 24 or more hours after a long-acting -agonist
* History of at least 1 asthma exacerbation leading to oral, IV or IM corticosteroid or ER/Urgent Care Center visit or hospitalization within the past year prior to Screening. This asthma exacerbation should not have been within 30 days prior to Screening
* Adequate cardiac, renal and hepatic function as determined by the principal investigator and demonstrated by Screening laboratory evaluations, questionnaires, and physical examination results that are within normal limits
* Subjects must be able to self-inject study medication or have a designee or healthcare professional who can inject the study medication

Exclusion Criteria:

* Active lung diseases (e.g., bronchitis, chronic obstructive pulmonary disease [COPD], interstitial lung disease, pulmonary fibrosis) other than asthma
* Current treatment for corticosteroid-resistant asthma (e.g., methotrexate [MTX], cyclosporine, gold salts, troleandomycin, immune globulin intravenous [IGIV], mycophenolate mofetil)
* History of cancer or lymphoproliferative disease other than a successfully and completely treated cutaneous squamous cell or basal cell carcinoma or carcinoma - in-situ of the cervix.
* History of listeria, human immunodeficiency virus (HIV), chronic or active Hepatitis B, an immunodeficiency syndrome, central nervous system (CNS) demyelinating disease or active TB
* Females who are pregnant or will not discontinue breast-feeding.
* Subject with a history of clinically significant drug or alcohol abuse in the last year
* Subjects with a poorly controlled medical condition.
* Abnormal, clinically significant screening laboratory and other analyses (including ECG).
* Subjects with any prior exposure to Tysabri® (natalizumab)
* Prior treatment with any TNF antagonist, including adalimumab

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2007-08

PRIMARY OUTCOMES:
The primary efficacy endpoint is the change from Baseline in post-bronchodilator FEV1 in subjects treated with adalimumab vs. placebo. | Week 16

SECONDARY OUTCOMES:
Proportion of subjects with at least one asthma exacerbation from Baseline to the end of the double-blind period | Week 16
Changes from Baseline in post-bronchodilator FEV1 | Time points other thanWeek 16
Change from Baseline in pre-bronchodilator FEV1
Change from Baseline (pre-bronchodilator) in FEV1 | 30 minutes postbronchodilator
Change from Baseline in percent predicted FEV1

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Paperiello, Study Director — Abbott